CLINICAL TRIAL: NCT07285239
Title: Randomized Phase 3 Trial of Belantamab Mafodotin or Daratumumab in Combination With Bortezomib, Lenalidomide and Dexamethasone for Newly Diagnosed Multiple Myeloma
Brief Title: Belantamab Mafodotin or Daratumumab With Bortezomib, Lenalidomide and Dexamethasone for Newly Diagnosed Multiple Myeloma
Acronym: PrE1005
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE1005; GSK 300057 (Other: GlaxoSmithKline)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed High-Risk Multiple Myeloma; Transplant Ineligible Multiple Myeloma; High-Risk Cytogenetic Multiple Myeloma; Belantamab Mafodotin; Daratumumab-Hyaluronidase; Daratumumab; Bortezomib; Lenalidomide; Decadron; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Bortezomib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Open-label, randomized (1:1) to either belantamab mafodotin or daratumumab given in combination with bortezomib, lenalidomide and dexamethasone (VRd) until progression. Participants will be stratified by IMWG risk criteria and intention to transplant at disease progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Belantamab Mafodotin (Experimental): Belantamab mafodotin in combination with bortezomib, lenalidomide and dexamethasone (VRd) until progression, unacceptable toxicity or participant withdrawal. 1 cycle = 28 days.
  Interventions: Drug: Arm A: Belantamab Mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Arm B: (Active Comparator): Daratumumab in combination with bortezomib, lenalidomide and dexamethasone (VRd) until progression, unacceptable toxicity or participant withdrawal. 1 cycle = 28 days.
  Interventions: Drug: Arm B: Daratumumab Hyaluronidase; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Arm A: Belantamab Mafodotin — 1.9 milligram/kilogram (mg/kg) intravenous (IV) will be administered every 8 weeks for first 24 weeks (Cycles 1-3), then 1.9 mg/kg every 12 weeks (Cycles 4+) until progression, unacceptable toxicity or participant withdrawal
  Other Names: GSK2857916; Blenrep; Belamaf
  Arms: Arm A: Belantamab Mafodotin
Drug: Arm B: Daratumumab Hyaluronidase — 1800 mg subcutaneous (SC) will be administered weekly from Week 1-8 (Cycles 1 and 2), every 2 weeks from Week 9-24 (Cycles 3-6), and every 4 weeks from Week 25 (Cycles 7+) onwards until progression, unacceptable toxicity or participant withdrawal
  Other Names: DARZALEX FASPRO™
  Arms: Arm B:
Drug: Bortezomib — 1.3 milligrams per square meter (mg /m²) SC on days 1, 8 and 15 of every 28 day bortezomib treatment cycle for 8 cycles
  Other Names: Velcade®
Drug: Lenalidomide — 25 mg orally (PO) Days 1-21 of every 28 day lenalidomide treatment cycle.
  Other Names: Revlimid®
Drug: Dexamethasone — 40 mg PO on Days 1, 8, 15, and 22 of each 28-day cycle
  Other Names: Decadron

SUMMARY:
Eligible participants with newly diagnosed myeloma who are not considered eligible for bone marrow transplant will be enrolled. Participants will be randomized to either belantamab mafodotin or daratumumab given in combination with bortezomib, lenalidomide and dexamethasone. Treatment will continue until disease progression, unacceptable side effects or withdrawal of consent.

Belantamab mafodotin is a targeted cancer treatment that works against multiple myeloma cells. It combines a homing device (an antibody) with a powerful cell-killing drug (a toxin), delivering the toxin directly to cancer cells while largely sparing healthy cells.

Minimal residual disease (MRD) testing will be done on bone marrow samples obtained standardly during your treatment. MRD shows whether a very small number of cancer cells can still be detected after treatment, even if standard lab tests shows no signs of cancer.

The purpose of this study is to evaluate if belantamab mafodotin, bortezomib, lenalidomide and dexamethasone (BVRd) improves minimal residual disease (MRD) negative status and/or prolongs progression-free survival (PFS) compared with daratumumab, bortezomib, lenalidomide and dexamethasone (DVRd) in participants with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This proposed Phase III multicenter, study is a randomized (1:1), open-label trial designed to show belantamab mafodotin in combination with bortezomib, lenalidomide and dexamethasone (VRd) will lead to higher minimal residual disease (MRD) negativity rate compared with daratumumab in combination with VRd in transplant ineligible newly diagnosed multiple myeloma (TI-NDMM). In addition, progression-free survival (PFS) will also be longer on the high-risk enriched population and the subgroup of high-risk cytogenetic participants.

After enrolling the first 400 patients, the study will limit accrual to patients with high risk NDMM to allow for enrichment of this subgroup of patients.

Belantamab mafodotin is a monoclonal antibody that targets B-cell maturation antigen (BCMA), a protein expressed on the surface of plasma cells, and releases a cytotoxic agent called Monomethyl auristatin F, which destroys the plasma cells.

International Myeloma Working Group (IMWG) criteria will be used for disease response.

MRD samples will be obtained on standard of care bone marrow procedures. MRD testing will be performed on samples at time of screening, suspected complete response (sCR), after confirmed CR at applicable time points from Cycle1, Day 1 at 6, 12, 18 (optional), 24, 30 (optional) and 36 months then annually until progression. MRD testing will not be performed in real-time for this study. Bone marrow samples will also be obtained for future research at screening and time of progression.

Research peripheral blood samples will be obtained to measure levels of belantamab mafodotin in the blood, immune responses or antibodies to belantamab mafodotin for patients receiving belantamab mafodotin. In addition, research blood samples will be obtained on all patients to measure soluble B-cell maturation antigen (sBCMA) to help diagnose, monitor treatment effectiveness, and predict the prognosis of multiple myeloma.

Patient-reported outcomes will also be performed.

ELIGIBILITY:
Eligibility Criteria:

* Patient must have suspected or confirmed newly diagnosed multiple myeloma (MM) by International Myeloma Working Group (IMWG) criteria and must not have received more than one cycle of any myeloma treatment.
* Patient must be considered ineligible for autologous stem cell transplantation by the treating physician, or willing to delay stem cell transplantation until first relapse or later.
* Patient must have measurable or evaluable disease as defined by having one or more of the following, obtained within 28 days prior to randomization.

  * ≥ 1g/dL monoclonal protein (M-protein) on serum protein electrophoresis
  * Involved free light chain ≥ 10 mg/dL or ≥ 100 mg/L AND abnormal serum immunoglobulin kappa to lambda free light chain ratio (<0.26 or >1.65)
  * ≥ 200 mg/24 hours of monoclonal protein on a 24-hour urine protein electrophoresis
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)
* Patient must be ≥ 18 years of age.
* Patient must have an Eastern Cooperative Group (ECOG) Performance Status (PS) of 0-2 (PS 3 allowed if secondary to pain).
* Patient must have the ability to understand and willingness to sign a written informed consent document.
* Patient must be willing to provide bone marrow (aspirate and/or biopsy) and blood samples for determination of International Myeloma Society (IMS) risk status and for research.
* Patient must have received no more than one cycle (28 days or less) of prior chemotherapy and no more than 160 mg of prior dexamethasone (or equivalent dose of prednisone) for treatment of symptomatic myeloma. Prior radiation therapy to symptomatic lesions is allowed provided there is no residual toxicity related to radiation and blood counts meet the study requirements.
* Patient must have a Serum Protein Electrophoresis (SPEP), Urine Protein Electrophoresis (UPEP), and serum Free Light Chain (FLC) assay performed within 28 days prior to registration. In addition, a bone marrow biopsy and/or aspirate is required within 28 days prior to registration if measurable disease is only present in bone marrow. Otherwise, a bone marrow examination must have been performed within 90 days prior to registration.
* Patient must have adequate organ function and marrow function as defined below, obtained ≤ 2 weeks prior to registration.

  * Absolute Neutrophil Count (ANC) ≥ 1000/microliter (mcL)
  * Platelets ˃75,000/mcL
  * Creatinine clearance (CrCl) ≥ 30 mL/min
  * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3x upper limit of normal (ULN)
  * Total Bilirubin ≤ 1.5x ULN or ≤ 3x ULN for patients with documented Gilbert's disease
* Patient must agree to register to the mandatory lenalidomide (Revlimid) Risk Evaluation and Mitigation Strategy (REMS) program and be willing and able to comply with the requirements of the REMS program.
* Patient must not be pregnant or breast-feeding due to the potential harm and teratogenic effects to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.
* Patient must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study, and for 3 months after the last dose of protocol treatment.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patient with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association (NYHA) Functional Classification. To be eligible for this trial, patient must be class 2 or better.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients must not have peripheral neuropathy ≥ Grade 2 on clinical examination or Grade 1 with pain at time of registration.
* Patients must not have any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Patient may have a history of current or previous deep vein thrombosis (DVT) or pulmonary embolism (PE) but must be willing to take some form of anti-coagulation as prophylaxis if they are not currently on full-dose anticoagulation.
* Patients must not have any known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients, or known sensitivity to mammalian-derived products.
* Patients must not have current corneal epithelial disease except mild punctuate keratopathy.
* Contact lenses are not allowed for participants while they are receiving belantamab mafodotin treatment.
* Patients must not have symptomatic amyloidosis or active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma-proliferative disorder, skin changes) at the time of screening.
* Patients must not receive any other concurrent chemotherapy, or any ancillary therapy considered investigational while on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2031-09 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
MRD Negative Status in All-Comers | 9 to 15 months
  MRD negative status, defined as achieving MRD negativity at 10^-5 sensitivity threshold assessed by next-generation sequencing (NGS) in patients achieving CR or better after 12 (+/- 3) months of treatment; MRD negativity is determined by the Adaptive Biotechnologies clonoSEQ® assay result; All-comers: the initial cohort of 400 consecutively enrolled patients, irrespective of IMS-IMWG risk status.
Progression-Free Survival (PFS) in High-Risk Cytogenetics Enriched Cohort | Up to 7 years
  PFS, defined as the time from the date of randomization to the date of first documented disease progression per IMWG criteria or death from any cause in the absence of progression, whichever occurs first; High-risk cytogenetics enriched cohort: includes the 400 all-comers and 100 additional patients with high-risk cytogenetics.

SECONDARY OUTCOMES:
PFS in High-Risk Cytogenetics Cohort | Up to 7 years
  PFS, defined as the time from the date of randomization to the date of first documented disease progression per IMWG criteria or death from any cause in the absence of progression, whichever occurs first; High-risk cytogenetics cohort: ~180 patients (~80 from all-comers and 100 from additional accrual) with high-risk cytogenetics.
Overall Survival (OS) | Up to 7 years
  OS, defined as the time from the date of randomization until the date of death due to any cause.
Best Response of Complete Response (CR) | Up to 7 years
  Defined as confirmed CR or better per IMWG criteria
Best Response of Very Good Partial Response (VGPR) | Up to 7 years
  Defined as confirmed VGPR, CR or better per IMWG criteria
Duration of Response (DoR) | Up to 7 years
  DoR, defined as the time from first documented evidence of partial response (PR) or better until progression (PD) or death due to PD (among participants who achieve confirmed PR or better)
Sustained MRD (sMRD) Negative Status | Up to 7 years
  sMRD, defined as achieving MRD negative status at 10-5 sensitivity threshold assessed by NGS at least twice, a minimum of 1 year apart and with no MRD positive result in between, during the time of confirmed CR or better response per IMWG criteria
Adverse Events (AEs) | While on study treatment and up to 70 days after the last dose of study medication
  Worst Grade 3 or Higher Treatment-Related Non-Hematologic and Overall Toxicity based on CTCAE v6.0
AEs Leading to Dose Modifications | While on study treatment and up to 70 days after the last dose of study medication
  AEs or Grade ≥ 2 Corneal Events Leading to Dose Modifications or Treatment Discontinuation
Corneal Events | While on study treatment and up to 70 days after the last dose of study medication
  Incidence of Grade ≥ 3 Corneal Events (Keratopathy Visual Acuity (KVA) scale)
Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 7 years
  Frequency and Score of Selected PRO-CTCAE Attributes
Health-Related Quality of Life (HRQoL) | Up to 7 years
  Change from Baseline in HRQoL as Measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and Functional Assessment of Cancer Therapy - Multiple Myeloma (FACT MM) Subscale

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, MD, Study Chair — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No
Data is proprietary